CLINICAL TRIAL: NCT01063088
Title: An Open Label, Phase 3 Study to Assess the Safety and Immunogenicity of a Vero Cell-Derived Trivalent Seasonal Influenza Vaccine, Strain Composition 2009/2010, in an Adult Population
Brief Title: Adult Safety Study of 2009/2010 Seasonal Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Gerald Aichinger, MD; Study Medical Director, Baxter Healthcare Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 720903; 2009-017781-23 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2010-07

CONDITIONS: Influenza
Keywords: Prophylaxis of seasonal influenza in adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccination (Experimental): Single 0.5 mL intramuscular injection of PreFluCel 2009/2010
  Interventions: Biological: Seasonal influenza vaccine (split virion, inactivated, prepared in Vero Cell cultures)

INTERVENTIONS:
Biological: Seasonal influenza vaccine (split virion, inactivated, prepared in Vero Cell cultures) — Single 0.5 mL intramuscular injection
  Other Names: PreFluCel 2009/2010

SUMMARY:
The purpose of the study is to verify the safety and immunogenicity of a trivalent seasonal influenza vaccine with strain composition according to World Health Organization (WHO)/European Union (EU) recommendation for the 2009/2010 season.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 59 years of age, inclusive, at the time of screening
* Subject has given written informed consent prior to study entry
* Subject is generally healthy, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination, such that the investigator would not hesitate to provide routine influenza immunization to the subject in the course of routine medical practice
* Subject agrees to keep a daily record of symptoms for the duration of the study
* If female of childbearing potential, subject presents with a negative urine pregnancy test immediately prior to vaccination on Study Day 1 and agrees to employ adequate birth control measures for the duration of the study
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subject has a history of severe allergic reaction or anaphylaxis
* Subject has an oral temperature of >= 37.5°C on the day of vaccination in this study Subject has a dermatologic condition or tattoos, which may interfere with injection site reaction rating
* Subject has received a live vaccine within 4 weeks or an inactivated or subunit vaccine within 2 weeks of study entry
* Subject has been vaccinated with seasonal influenza vaccine for the 2009/2010 season
* Subject currently has or had a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder
* Subject has any inherited or acquired immunodeficiency
* Subject has a disease or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (> 800 μg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs.
* Subject has a functional or surgical asplenia
* Subject has a known or suspected problem with alcohol or drug abuse
* Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie., children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.
* If female, subject is pregnant or lactating at the time of study enrollment
* Subject has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a trivalent seasonal influenza vaccine with strain composition according to WHO/EU recommendation for the 2009/2010 season in an adult population through the first seven post vaccination days | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Aichinger, MD, Study Director — Baxter Healthcare Corporation
Locations (2):
- Sanatorium Leech, Graz, Austria
- ZU Gent, Centrum voor vaccinologie, Ghent, Belgium